CLINICAL TRIAL: NCT03629717
Title: RANKL Inhibition and Breast Tissue Biomarkers in Premenopausal Women With Dense Breasts
Brief Title: RANKL Inhibition and Breast Tissue Biomarkers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201801105
Record Dates: First submitted 2018-08-01; First posted 2018-08-14 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Prevention; Mammographic Density
Keywords: Mammographic density; Premenopausal; Breast cancer; Chemoprevention; Denosumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Denosumab; Blood Specimen Collection; Calcium; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Denosumab (Experimental): An ultrasound-guided core needle breast biopsy will be performed on day 1 prior to the intervention. A single dose of subcutaneous denosumab 60mg will be administered immediately after the core biopsy on day 1. This will take place on an outpatient basis. Repeat core-needle biopsy will take place on Day 60 (+/-10 days). Blood samples will also be collected at the time of core-needle biopsy to allow for biomarker assay. Gene expression analyses will be done using NanoString nCounter gene expression system.
  Interventions: Procedure: Ultrasound-guided core needle biopsy; Drug: Denosumab; Procedure: Blood draw; Drug: Calcium; Drug: Vitamin D

INTERVENTIONS:
Procedure: Ultrasound-guided core needle biopsy — Tissue collection for this research proposal will be used for research purposes only and will not inform participant care
Drug: Denosumab — Denosumab is a human IgG2 monoclonal antibody with affinity and specificity for human RANKL
  Other Names: Xgeva; Prolia
Procedure: Blood draw — 20 mL of fasting whole blood will be collected before denosumab (Day 1) and one month after denosumab administration (day 60 +/- 10 days)
Drug: Calcium — 1200mg daily
Drug: Vitamin D — 800 IU daily

SUMMARY:
A robust knowledge of how to reduce breast density could play a key role in breast cancer prevention in premenopausal women, but viable preventative targets to reduce breast density-associated breast cancer risk are yet to be developed. The investigators propose to investigate the effect of RANKL inhibition with denosumab on breast tissue markers in high-risk premenopausal women with dense breasts. Study findings could provide robust evidence to move forward with a clinical trial targeting RANKL inhibition in premenopausal breast cancer prevention.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Premenopausal.
* At least 35 years of age.
* Dense breasts on routine mammogram.
* Willing to take calcium (1,200mg) and vitamin D (800 IU) daily.
* At increased risk for breast cancer using any of the following:

  * Positive family history of breast cancer
  * Breast cancer risk prediction models
* Able and willing to return for repeat biopsy.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Current use of tamoxifen, aromatase inhibitors, or bisphosphonates.
* Concurrently participating in another cancer chemoprevention trial (unless no longer receiving the intervention).
* Pregnant or lactating.
* Recent tooth extraction or dental procedure.
* Unhealed and/or planned dental/oral surgery.
* History of osteonecrosis/osteomyelitis of the jaw.
* History of osteoporosis or severe osteopenia.
* Unable/unwilling to return for repeat biopsy.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Effect of denosumab on breast tissue gene pathway gene expression | Between baseline and day 60
  The investigators will evaluate changes in pathway gene expression between baseline and day 60 using NanoString NCounter platform
Effect of denosumab on pathways that may influence breast cancer development as measured by spatial transcriptomic analysis | Between baseline and day 60
  The investigators will evaluate changes in breast tissue spatial transcriptomics.
Effect of denosumab on pathways that may influence breast cancer development as measured by metabolomic analysis | Between baseline and day 60
  The investigators will evaluate changes in metabolomics.

SECONDARY OUTCOMES:
Correlation of breast tissue gene expression with circulating biomarker levels | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Adetunji T Toriola, M.D., Ph.D., MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu